CLINICAL TRIAL: NCT05940571
Title: Phase I/Ib Trial of Single Agent MBF-362 in Solid Tumors
Brief Title: First Phase Clinical Trial of Single Agent MBF-362 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medibiofarma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MBF-362CT-01; 2022-001154-30 (EudraCT Number)
Record Dates: First submitted 2023-06-30; First posted 2023-07-11 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Cancer; solid tumors; Prostaglandin E receptor; immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- MBF-362 128.7 mg (Experimental): Drug: One MBF-362 128.7 mg hard gelatin capsule EP2/EP4 antagonist 28 days single oral daily dosing cycles
  Interventions: Drug: MBF-362
- MBF-362 257.4 mg (Experimental): Drug: Two MBF-362 128.7 mg hard gelatin capsules EP2/EP4 antagonist 28 days single oral daily dosing cycles
  Interventions: Drug: MBF-362
- MBF-362 514.8 mg (Experimental): Drug: Four MBF-362 128.7 mg hard gelatin capsules EP2/EP4 antagonist 28 days single oral daily dosing cycles
  Interventions: Drug: MBF-362
- MBF-362 772.2 mg (Experimental): Drug: Six MBF-362 128.7 mg hard gelatin capsule EP2/EP4 antagonist 28 days single oral daily dosing cycles
  Interventions: Drug: MBF-362

INTERVENTIONS:
Drug: MBF-362 — Drug: One MBF-362 128.7 mg hard gelatin capsule EP2/EP4 antagonist 28 days single oral daily dosing cycles

SUMMARY:
This is an open, single center Phase Iclinical trial to evaluate the safety, tolerability, and preliminary efficacy of MBF-362 in patients with solid tumors.

DETAILED DESCRIPTION:
The phase I dose escalation will be conducted utilizing the standard 3+3 dose escalation method. Pharmacokinetic (PK) data will be obtained for MBF-362.

The phase I dose expansion will consist of 1 group including solid tumors cancer patients. Pharmacodynamic (PD) data will be obtained for potential biomarker analysis with pre-treatment and on-treatment tumor biopsies.

Phase I Dose Escalation (3+3 Design): the MTD will be defined as the highest dose level at which less than 2 out of 6 patients (<33%) experience DLT in Cycle 1 (first 28 days).

Phase I Safety Expansion once RP2D has been declared for MBF-362 using the standard 3+3 design, up to 20 additional solid tumor cancer patients may be treated at the RP2D to further explore safety and tolerability of the selected MBF-362 dose.

Patients must have histologically or cytologically confirmed cancer with at least one measurable lesion, with adequate organ and marrow function, and with ECOG performance status of 0-1. Eligible patients must have received at least one prior line of therapy for their disease.

ELIGIBILITY:
Inclusion Criteria:

* These criteria are similarly applicable to patients enrolled to the phase I dose escalation and to the phase IB dose expansion portions of the trial.

  1. Advanced/metastatic histologically confirmed solid tumor. All types of solid tumors are allowed in the study
  2. At least 1 measurable lesion per Response Evaluation Criteria in solid tumor (RECIST 1.1).
  3. Patients who have progressed to the standard therapy and have no approved optional therapy available.
  4. ECOG performance status of 0/1
  5. Age greater than 18 years (inclusive).
  6. Adequate bone marrow, renal and hepatic function
  7. Able and willing to give valid written consent for available archival tumor samples (mandatory) and tumor biopsies before and during protocol (immune)therapy (optional in escalation phase and mandatory in expansion phase).
  8. Prior immunotherapy is also allowed.

Exclusion Criteria:

* These criteria are similarly applicable to patients enrolled to the phase I dose escalation and to the phase IB dose expansion portions of the trial.

  1. Participation in another clinical study with an investigational product during the last 4 weeks or 5 half-lives prior to starting on treatment.
  2. Symptomatic and/or untreated Brain Metastases
  3. Pregnancy or breast feeding
  4. Serious uncontrolled medical disorder or active infection that in the investigator's opinion would impair the patient's ability to receive study treatment.
  5. Concurrent use of other anticancer approved or investigational agents is not allowed.
  6. Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
  7. Prior malignancy in past 2 years or as identified in Section 7.2 of this protocol.
  8. Patients receiving oral or systemic steroids 2 weeks prior to dosing with MBF-362
  9. Patients receiving >4 doses of anti-inflammatory (NSAID) treatments, modulators of the COX-2 pathway or aspirin 1 week prior to dosing with MBF-362
  10. Patients with a history of gastric/duodenal ulcers, colitis and/or gastrointestinal bleeding, severe gastrointestinal adverse reactions
  11. Patients with a history of anaphylaxis, uncontrolled asthma or allergy/hypersensitivity/intolerance to NSAIDs, COX-2 inhibitors or aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events | 28 Days
  AEs will be described by system organ class and preferred tem using the Medical Dictionary for Regulatory Activities (MedDRA)
The Maximun Tolerated Dose (MTD) of MBF-362 | 28 Days
  The MTD evaluation will be based on the DLT Evaluable Population which includes all patients enrolled in the dose-escalation portion of the trial, who receive the protocol-assigned treatment with MBF-362 and complete the safety follow-up through the DLT evaluation period or experience a DLT during the DLT evaluation period

SECONDARY OUTCOMES:
Time to MBF-251 peak concentration in plasma "Tmax" | Between day 1 and 2, and day 8 and 9 of cycle 1, and between day 1 and 2 of cycle 2 (each cycle is 28 days)
  The parameter will be calculated from plasma samples collected at days 1, day 2, day 8 and day 9 after drug administration for cycle 1, and at days 1 and 2 for cycle 2. It will consist in the time (in minutes) to reach the maximum "MBF-251" concentration in plasma samples of patients after oral administration of MBF-362
MBF-251 peak concentration in plasma "Cmax" | Between day 1 and 2, and day 8 and 9 of cycle 1, and between day 1 and 2 of cycle 2 (each cycle is 28 days)
  The parameter will be calculated from plasma samples collected at days 1, day 2, day 8 and day 9 after drug administration for cycle 1, and at days 1 and 2 for cycle 2. It will consist in the time (in minutes) to reach the maximum "MBF-251" concentration in plasma samples of patients after oral administration of MBF-362
The area under MBF-251 plasma concentration-time curve to infinite time "AUC(0-inf) | Between day 1 and 2, and day 8 and 9 of cycle 1, and between day 1 and 2 of cycle 2 (each cycle is 28 days)
  The parameter will be calculated from plasma samples collected at days 1, day 2, day 8 and day 9 after drug administration for cycle 1, and at days 1 and 2 for cycle 2. It will consist in the area under the concentration-time curve from zero up to ∞ with extrapolation of the terminal phase. "AUC(0-inf)" will be given in Amount·time/ volume units
MBF-251 half-life in plasma " t½" | Between day 1 and 2, and day 8 and 9 of cycle 1, and between day 1 and 2 of cycle 2 (each cycle is 28 days)
  The parameter will be calculated from plasma samples collected at days 1, day 2, day 8 and day 9 after drug administration for cycle 1, and at days 1 and 2 for cycle 2. It will consist in the terminal half-life of PBF-251 in plasma. "t½" will be given in hours (h)
Efficacy of MBF-362 treatment as measured by Objective response rate (ORR) | 2 years
  ORR: Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).ORR is defined as confirmed complete response (CR) or partial response (PR) based on modified RECIST v1.1.
Efficacy of MBF-362 treatment as measured by Disease control rate (DCR) | 2 years
  The disease control rate (DCR) will be estimated considering the following variables: Complete response (CR), Partial response (PR) and stable disease (SD) as described by Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). These variables will be assessed based on Imaging-based evaluation methods as chest x-ray, conventional computed tomography (CT) and magnetic resonance imaging (MRI).
Efficacy of MBF-362 treatment as measured by duration of response (DoR) | 2 years
  Duration of response (DoR) is defined as the duration from the first documentation of OR to the first documented disease progression or death due to any cause, whichever occurs first.
Efficacy of MBF-362 treatment as measured by progression-free survival (PFS) | 2 years
  Progression-free survival (PFS) will be measured from the start of treatment until the documentation of disease progression or death due to any cause, whichever occurs first. For subjects who are alive and progression-free at the time of data cut-off for analysis, PFS will be censored at the last tumor assessment date.
Efficacy of MBF-362 treatment as measured by overall survival (OS) | 2 years
  Overall survival (OS) will be determined as the time from the start of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Catalan de Oncología, L'Hospitalet de Llobregat, Barcelona, Spain